CLINICAL TRIAL: NCT02855307
Title: A Single-blind, Randomized, Cross-over Study to Assess the Efficacy of Single-hormone Closed-loop Strategy at Preventing Hypoglycemia During Unannounced and Announced Exercise in Adults With Type 1 Diabetes
Brief Title: Closed-loop Control of Glucose Levels (Artificial Pancreas) During Postprandial Exercise in Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLASS-16
Record Dates: First submitted 2016-08-01; First posted 2016-08-04 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Type 1 Diabetes
Keywords: Closed-loop system; Artificial pancreas; Exercise; Hypoglycemia; Insulin; Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia; Insulin Resistance | interventions — Exercise; Insulin Infusion Systems; Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Unannounced exercise (Active Comparator): The target blood glucose of the algorithm will be as usual. A pre-meal full insulin bolus will be given.
  Interventions: Other: 60-minute exercise; Device: Insulin pump; Device: Dexcom G4 Platinum glucose sensor; Drug: Insulin; Other: Single-hormone closed-loop strategy
- Announced exercise with pre-meal full bolus (Active Comparator): The target blood glucose of the algorithm will be increased and a pre-meal full bolus will be given
  Interventions: Other: 60-minute exercise; Device: Insulin pump; Device: Dexcom G4 Platinum glucose sensor; Drug: Insulin; Other: Single-hormone closed-loop strategy
- Announced exercise with reduced insulin bolus (Active Comparator): The target blood glucose of the algorithm will be increased and the pre-meal insulin bolus will be reduced by 33%.
  Interventions: Other: 60-minute exercise; Device: Insulin pump; Device: Dexcom G4 Platinum glucose sensor; Drug: Insulin; Other: Single-hormone closed-loop strategy

INTERVENTIONS:
Other: 60-minute exercise — Patients will be admitted at the research clinical facility at 6:30. The artificial pancreas intervention will start at 7:00. A standardized breakfast will be served at 8:00. At 9:30, patients will performed a 60-minute exercise on the ergocycle at 60% of VO2 max. At 11:30, patients will be switched to standard insulin pump therapy and a lunch will be served. Patients will be discharged after lunch consumption.
Device: Insulin pump — Patient's insulin pump will be used to infuse insulin.
Device: Dexcom G4 Platinum glucose sensor — The Dexcom G4 Platinum glucose sensor will be used to measure glucose levels.
Drug: Insulin — Patient's usual fast-acting insulin analog will be used.
Other: Single-hormone closed-loop strategy — Variable subcutaneous insulin infusion rates will be used to regulate glucose levels. Patient's usual fast acting insulin analog (Lispro, Aspart or Guilisine) will be infused using the patient's pump. The glucose level as measured by the real time sensor (Dexcom G4 Platinum, Dexcom Inc.) will be entered manually into the computer every 10 minutes. The pump's infusion rate will then be changed manually based on the computer generated recommendation infusion rates.

SUMMARY:
Regular physical activity is associated with many health benefits for individuals with type 1 diabetes including improved cardiovascular fitness and vascular health, decreased insulin requirements, improved body composition and quality of life. However, exercise-induced hypoglycemia is very frequent and thus is the main limiting factor for physical activity practice in this population.

The artificial pancreas is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings. The artificial pancreas has the potential to reduce the risk of exercise-induced hypoglycemia but the importance of announcing exercise to the artificial pancreas is yet to be explored.

The objective of this study is to investigate 1) if announcing postprandial exercise to the artificial pancreas is beneficial in reducing the risk of hypoglycemia and 2) if an insulin bolus reduction is necessary when announcing the exercise to the artificial pancreas.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of old.
2. Clinical diagnosis of type 1 diabetes for at least one year.
3. The subject will have been on insulin pump therapy for at least 3 months.
4. Last (less than 3 months) HbA1c ≤ 12%.

Exclusion Criteria:

1. Clinically significant microvascular complications: nephropathy (estimated glomerular filtration rate below 40 ml/min), neuropathy (especially diagnosed gastroparesis) or severe proliferative retinopathy as judged by the investigator.
2. Recent (< 3 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. Use of medication with an effect on heart rate (e.g. beta-blockers).
4. Abnormal blood panel and/or anemia.
5. Ongoing or planned pregnancy.
6. Severe hypoglycemic episode within two weeks of screening.
7. Other serious medical illness likely to interfere with study participation or with the ability to complete the exercise periods by the judgment of the investigator (e.g. orthopedic limitation).
8. Failure to comply with team's recommendations (e.g. not willing to eat snack, not willing to change pump parameters, etc).
9. Problems with venous access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-09; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Percentage of time of plasma glucose levels spent below 3.9 mmol/L | From 9:30 to 11:30 (120 minutes)

SECONDARY OUTCOMES:
Relative decrease in glucose levels during exercise compared to pre-breakfast levels | From 8:00 to 10:50 (170 minutes)
  Difference between pre-breakfast levels and the lowest glucose level from the start of the exercise until 20 minutes after exercise
Number of patients experiencing exercise-induced hypoglycemia requiring treatment | From 9:30 to 10:30 (60 minutes)
Decremental area under the curve from the start of the exercise | From 9:30 to 11:00 (90 minutes)
Percentage of time of plasma glucose levels spent below 3.9 mmol/L | From 9:30 to 10:30 (60 minutes)
Percentage of time of plasma glucose levels spent below 3.3 mmol/L | From 9:30 to 10:30 (60 minutes)
Percentage of time of plasma glucose levels spent below 2.8 mmol/L | From 9:30 to 10:30 (60 minutes)
Percentage of time of plasma glucose levels spent between 3.9 and 7.8 mmol/L | From 9:30 to 10:30 (60 minutes)
Percentage of time of plasma glucose levels spent above 10 mmol/L | From 9:30 to 10:30 (60 minutes)
Percentage of time of plasma glucose levels spent above 13.9 mmol/L | From 9:30 to 10:30 (60 minutes)
Percentage of time of plasma glucose levels spent above 16.7 mmol/L | From 9:30 to 10:30 (60 minutes)
Mean plasma glucose levels | From 8:00 to 11:30 (210 minutes)
Standard deviation of glucose levels | From 8:00 to 11:30 (210 minutes)
Coefficient of variation of glucose levels | From 8:00 to 11:30 (210 minutes)
Mean time (minutes) to the first hypoglycemic event | From 9:30 to 10:30 (60 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tagougui S, Taleb N, Legault L, Suppere C, Messier V, Boukabous I, Shohoudi A, Ladouceur M, Rabasa-Lhoret R. A single-blind, randomised, crossover study to reduce hypoglycaemia risk during postprandial exercise with closed-loop insulin delivery in adults with type 1 diabetes: announced (with or without bolus reduction) vs unannounced exercise strategies. Diabetologia. 2020 Nov;63(11):2282-2291. doi: 10.1007/s00125-020-05244-y. Epub 2020 Aug 1. PMID 32740723